CLINICAL TRIAL: NCT06145048
Title: A Phase 2, Multi-center, Open-label Study to Evaluate the Safety and Efficacy of VGT-309, a Tumor-Targeted, Activatable Fluorescent Imaging Agent, in Subjects Undergoing Surgery for Cancer in the Lung
Brief Title: Phase 2B Safety and Efficacy Study of VGT-309 in Subjects With Cancer in the Lung.
Acronym: VISUALIZE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vergent Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGT-309-2B-2023
Record Dates: First submitted 2023-11-13; First posted 2023-11-22 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer; Lung Metastases
Keywords: Lung Cancer; Metastatic Cancer in Lung
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is an open label study in which all subjects will receive a dose of 0.32mg/kg VGT-309 (based on their weight) at 12-36 hours pre-surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 0.32 mg/kg VGT-309 (Experimental): 0.32 mg/kg VGT-309 given over 15-20 minutes by syringe pump
  Interventions: Drug: VGT-309

INTERVENTIONS:
Drug: VGT-309 — Intravenous drug to be given over 15-20 minutes by syringe pump.

SUMMARY:
This is a Phase 2, multi-center, open-label study to evaluate the safety and efficacy of VGT-309, a tumor-targeted, activatable fluorescent imaging agent, in subjects undergoing surgery for proven or suspected cancer in the lung. Approximately 100 subjects will be enrolled to ensure at least 86 subjects are evaluable with the option to expand enrollment by protocol amendment if deemed necessary by the DSC to meet primary and/or secondary objectives.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, open-label study to evaluate the safety and efficacy of VGT-309, a tumor-targeted, activatable fluorescent imaging agent, in subjects undergoing surgery for proven or suspected cancer in the lung. Approximately 100 subjects will be enrolled to ensure at least 86 subjects are evaluable with the option to expand enrollment by protocol amendment if deemed necessary by the DSC to meet primary and/or secondary objectives.

Following agreement with and signing of the informed consent, subjects will undergo screening measurements for the study within 4 weeks prior to the anticipated dosing:

1. Medical, surgical and medication history.
2. Complete physical exam, including vital signs and height
3. Weight (needed for dose calculation)
4. Chemistry, hematology, coagulation and urinalysis with microscopy clinical laboratory studies.
5. 12-lead ECG.
6. Serum pregnancy test for females of child-bearing potential.

After meeting all enrollment criteria, each subject will receive 0.32 mg/kg VGT-309 by IV administration 12-36 hours prior to surgery (refer to section VGT-309 Dosing, below). Subjects will be observed for 1 hour after dosing is completed and asked about possible treatment emergent adverse events.

Subjects will undergo surgical resection within 12-36 hours after completion of VGT-309 dosing. Measurements of efficacy will be taken during surgery and during the pathological examination of all surgical specimens. (Refer to Efficacy Endpoints and Efficacy Assessments sections).

Following surgery, subjects will be monitored for safety during their hospitalization. Between 7 to 14 and 25 to 35 days after surgery, the subjects will return to the clinic or have a telehealth visit for final safety assessments. At the last visit, if there are no adverse events requiring further follow up, subjects will then be released from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to sign the informed consent and comply with study procedures.
2. Be at least 18 years of age.
3. Meet the following conditions:

   Female participants must be of non-childbearing potential, or, If of childbearing potential, be non-pregnant or non-lactating and agree to use highly effective contraception from screening through Day 30 after treatment.

   Male participants, if not surgically sterilized, and if engaging in sexual intercourse with a female partner of childbearing potential, must be willing to use highly effective contraception from screening through 30 days after treatment and agree not to donate semen during this waiting period.

   Highly effective contraception involves the use of a condom for the male, plus one of the following for the female:

   Oral, injectable, implantable, intravaginal, or transdermal hormonal contraceptives, or Intrauterine device or intrauterine hormone-releasing system NOTE: Subjects who abstain from heterosexual intercourse as their usual and preferred lifestyle, will not be required to use contraception as described above. They are required to maintain abstinence from screening through Day 30 after treatment.

   Note: Subjects in a same sex relationship, must use a barrier form of contraception (e.g., condom, diaphragm) to protect against the transfer of the study drug in any bodily fluids.
4. Have a lung nodule or mass that might be considered primary lung cancer or lung metastases whether or not it is biopsy-proven before surgery.
5. Be scheduled to undergo standard of care surgical resection for a lung nodule or mass with diagnostic and/or curative intent
6. Have acceptable kidney and liver functions at study entry as evidenced by:

ALT/AST < 1.5 times the upper limit of normal Calculated Creatinine Clearance (CrCl) ≥ 50 ml/min Total bilirubin < 1.5 times the upper limit of normal Have an ECOG score of 0-2. Meet all standard of care surgical and general anesthesia requirements. 7) Have not participated in an interventional clinical trial within the last 30 days.

-

Exclusion Criteria:

1. Not a candidate for standard of care surgery based on opinion of the surgeon, anesthesiologist, or other consulting physician.
2. Have a known allergy or reaction to ICG, other radiographic contrast agent, or any component of VGT-309.
3. Have congenital long QT syndrome or QTcF > 470ms by history or at Screening ECG.
4. Prisoners, institutionalized individuals, or are unable to consent for themselves.
5. Have any other co-morbidity or habit that the Investigator believes will interfere with their ability to comply with and complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Measurements taken under SOC surgical procedures and under NIR imaging | During surgery and up to 1 month post-surgery
  Proportion of subjects with at least one Clinically Significant Event (CSE) defined as:
  A. Intraoperative localization of one or more preoperatively identified lung lesions using VGT-309 with NIR imaging B. Identification of one or more synchronous or occult lung lesions using VGT-309 with NIR imaging when standard surgical techniques using white light and palpation and preoperative imaging failed to identify the lesion(s C. Identification of fluorescence within ≤10 mm from the inside edge of the closest staple line as measured by the investigator ex vivo in the operating room using NIR imaging, with pathologic margin confirmed by histologic examination to be ≤ 10 mm.
  D. Identification of lymph nodes by VGT-309 with NIR imaging confirmed by histologic examination to be cancerous.

SECONDARY OUTCOMES:
Measurements taken under SOC surgical procedures and under NIR imaging | During surgery and up to one month post-surgery
  Efficacy: To evaluate the sensitivity, positive predictive value (PPV), and 1-PPV of VGT-309 with NIR imaging for lesion(s) in vivo. Definitions to apply:
  1. Sensitivity is defined as the probability that the tissue fluoresces when it is cancer, as confirmed by histology (TP/(TP+FN)) *
  2. Positive predictive value (PPV) is defined as the probability that a tissue sample contains cancer on histologic exam if it fluoresces ((TP/(TP+FP))
  3. 1-Positive predictive value (1-PPV) is defined as the probability that a tissue sample does not contain cancer when it fluoresces ((FP/(TP+FP))* Where: * TP = true positive, FP = false positive, FN = false negative

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Scribner, MD, Study Director — Vergent Bioscience
Locations (6):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - Orlando Health Cancer Institute, Orlando, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- St. Vincent's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
The joint publication will be coordinated by Vergent. There is no need for individual sites to review specific IPD from other sites.